CLINICAL TRIAL: NCT01770483
Title: The Role Of Nitazoxanide, Interferon Alfa And Ribavirin In Treatment Of Hepatitis C Infected Type 2 Diabetic Patients
Acronym: HEP-C-FM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Collaborators: Getz Pharma (Industry)
Responsible Party: Principal Investigator, Prof. Faisal Masud, Principal SIMS, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMS
Record Dates: First submitted 2013-01-08; First posted 2013-01-17 (Estimated); Results first posted 2013-04-17 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Hepatitis C, Chronic; DIABETES MELLITUS Type 2
Keywords: Nitazoxanide,; Sustained viral response; Type 2 DIABETICS
MeSH Terms: conditions — Hepatitis C, Chronic; Diabetes Mellitus, Type 2 | interventions — nitazoxanide; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Tablet Nitazoxanide 500mg twice daily will be added to the injection conventional interferon alfa 3 Million International Units alternate days and capsule Ribavirin 400mg-1200mg weekly for six months
  Interventions: Drug: nitazoxanide; Drug: conventional interferon alfa; Drug: Ribavirin
- control group (Active Comparator): Injection conventional interferon alfa 3 Million International Units alternate days and capsule ribavirin 400mg-1200mg weekly for six months
  Interventions: Drug: conventional interferon alfa; Drug: Ribavirin

INTERVENTIONS:
Drug: nitazoxanide — nitazoxanide 500mg twice daily
  Other Names: tablet nizonide500mg; tablet atizox500mg
  Arms: study group
Drug: conventional interferon alfa — Inj interferon 3 Million International Units thrice weekly
  Other Names: Inj uniferon 3 Million International Units
Drug: Ribavirin — ribazole
  Other Names: Ribavirin 400mg-1200mg

SUMMARY:
The purpose of this study is to investigate if nitazoxanide used in combination with interferon alfa and ribavirin is effective in treating Hepatitis c infected type 2 Diabetic patients by improving their sustained viral response by more than 80%.Considering that the study is being conducted in a third world country like Pakistan, the standard treatment of hepatitis C is not cost effective. The aim is to introduce a new treatment comparable in efficacy to peginterferon and also cost effective.

DETAILED DESCRIPTION:
After taking proper informed consent from patients, patients who fulfill the research criteria are randomized into 2 groups (control/study). Patients in both groups will be treated with conventional interferon alfa and Ribavirin.Those in study group will be given tab nitazoxanide 500mg twice daily in addition to conventional treatment. The patients will be followed up at regular intervals: 0,4,12,24,48 week.At each visit Hepatitis C Virus(PCR)RNA, Liver function tests, complete blood count will be done.

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis C genotype 3a
* Hepatitis C Virus(PCR)RNA Detected
* Alanine transaminase >60
* Diabetic HbA1c<8
* BMI>23

Exclusion Criteria:

* Previously treated Hepatitis C patients
* Pregnant females
* Decompensated liver disease,Child class B OR above
* Thyroid disease,Thyroid stimulating hormone>10,0.05
* Absolute neutrophil count<1500,Platelets<80,000,Hb<10g Female,<11g Male
* Severe cardiac disease,New York Heart Association2
* Moderate to severe depression assessed by Beck Depression Inventory scale

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2011-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: FAISAL MASUD, FRCP, Study Director — Principal SIMS/Services hospital lahore; AMENA MIRZA, MRCP,FCPS, Principal Investigator — Senior registrar ,Services hospital lahore/SIMS; Madiha Fida, MBBS, Principal Investigator — House Officer Services Hospital Lahore
Locations (1):
- Endocrinology and Diabetes management centre, Lahore, Punjab Province, Pakistan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data was collected from diabetic patients coming to diabetes management center Services Hospital Lahore. Recruitment started on july 2011 and last patient was recruited in March 2012.
Pre-assignment Details: Initially 153 patients were recruited but only 66 patients were enrolled in the trial based on our inclusion criteria. Following patients were excluded:
  * 33 because of HCV genotype other than 3
  * 18 because of normal ALT
  * 9 with undetectable HCV PCR
  * 2 because of thyroid dysfunction
  * 25 were lost to follow up
Groups:
- Control Group: Injection conventional interferon alfa 3 Million International Units alternate days and capsule ribavirin 400mg-1200mg weekly for six months
  Ribavirin : ribazole
  conventional interferon alfa : Inj interferon 3 Million International Units thrice weekly
- Study Group: Tablet Nitazoxanide 500mg twice daily will be added to the injection conventional interferon alfa 3 Million International Units alternate days and capsule Ribavirin 400mg-1200mg weekly for six months
  Ribavirin : ribazole
  nitazoxanide : nitazoxanide 500mg twice daily
  conventional interferon alfa : Inj interferon 3 Million International Units thrice weekly
Period: Overall Study
Arm/Group | Control Group | Study Group
Started | 33 | 33
Completed | 33 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Study Group | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.30 (6.07) | 47.21 (5.464) | 47.26 (5.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 18 | 19 | 37
Region of Enrollment [Number; unit: participants]
  Pakistan | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Sustained Viral Response,
Description: Sustained viral response ,is negative Hepatitis C Virus(PCR)RNA test six months after end of treatment.
Time Frame: 48 WEEK
Population: Sample size has been calculated using Epi-Info 3.5.1 with the following assumptions.
  Reported ETR with Interferon + Ribavarin = 44 % Expected ETR with Interferon + Ribavarin + Nitazoxanide = 80 % Confidence Level = 95 % Power of Study = 80% Calculated Sample Size = 66 i.e. 33 in each group.
Measure: Number; unit: participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 33 | 33
participants | 13 | 11

2. Secondary Outcome: Normalization of Alanine Transferase Test
Description: Liver function test,showing resolution of the inflammation of liver parenchyma
Time Frame: 48week
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Control Group | Study Group
Number analyzed (Participants) | 33 | 33
participants | 11 | 11

ADVERSE EVENTS:
Time Frame: 1 year and 8 months
Arm/Group | Control Group | Study Group
Serious Adverse Events (participants affected / at risk) | 2/33 | 3/33
Other Adverse Events (participants affected / at risk) | 33/33 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=33) | Study Group (N=33)
hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
diabetic foot (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=33) | Study Group (N=33)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Flu (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 29 (29)
Dry Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 16 (16) | 23 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No